CLINICAL TRIAL: NCT06378359
Title: Effectiveness of Screening and Decolonization of S. Aureus to Prevent S. Aureus Surgical Site Infections in Surgery Outpatients
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: IDIM-2023-32364
Record Dates: First submitted 2024-04-18; First posted 2024-04-22 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Staphylococcus Aureus Colonization; Surgical Site Infections; Healthcare Associated Infections
MeSH Terms: conditions — Surgical Wound Infection; Cross Infection | interventions — Mass Screening; Ethanol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Arm 1a: screening for SA carriage and using the three-drug decolonization bundle among patients with SA colonization
  Interventions: Other: Screening and decolonization for SA carriers with the 3 drug bundle
- Arm 1b: non SA carriers in this arm will get two pre-op showers with an antiseptic soap
  Interventions: Other: No screening for SA
- Arm 2: giving pre-surgical patients the three drug decolonization bundle without screening.
  Nasal mupirocin, chlorhexidine gluconate (CHG) mouth rinse, and CHG body wash
  Interventions: Other: no screening
- Arm 3: giving pre-op nasal povidone iodine without screening
  Interventions: Other: Nasal povidone-iodine on surgery day plus 2 CHG pre-op showers without screening.
- Arm 4: giving nasal alcohol gel without screening
  Interventions: Other: Nasal alcohol gel on surgery day plus 2 CHG pre-op showers without screening

INTERVENTIONS:
Other: Screening and decolonization for SA carriers with the 3 drug bundle — nasal mupirocin, chlorhexidine gluconate (CHG) mouth rinse and CHG soap showers x 5 days and non-SA carriers receive 2 CHG pre-op showers
  Groups: Arm 1a
Other: No screening for SA — All receive the 3 drug bundle, Nasal mupirocin, chlorhexidine gluconate (CHG) mouth rinse, and CHG body wash
  Groups: Arm 1b
Other: no screening — giving pre-surgical patients the three drug decolonization bundle without screening
  Groups: Arm 2
Other: Nasal povidone-iodine on surgery day plus 2 CHG pre-op showers without screening. — Nasal povidone-iodine on surgery day plus 2 CHG pre-op showers without screening.
  Groups: Arm 3
Other: Nasal alcohol gel on surgery day plus 2 CHG pre-op showers without screening — Nasal alcohol gel on surgery day plus 2 CHG pre-op showers without screening
  Groups: Arm 4

SUMMARY:
The purpose of the study is to determine the effectiveness, safety, and health-care utilization and costs of a preoperative Staphylococcus aureus (SA) screening and decolonization bundle, (5 days of nasal mupirocin ointment, chlorhexidine gluconate (CHG) body wash, and CHG mouth rinse), in eradicating SA carriage compared to other SA decolonization approaches. The study will conduct a single center pilot trial to compare efficacy of different SA decolonization approaches in pre-surgical patients, in eradicating SA carriage, after obtaining informed consent.

The study will compare four different approaches, Arm 1) screen for SA carriage and using the three-drug decolonization bundle for 5 days among patients with SA colonization, non SA carriers in this arm will get two pre-op showers with CHG soap, Arm 2) all participants receive the three drug decolonization bundle, Arm 3) all receive pre-op nasal povidone iodine the day of surgery plus two pre-op showers with CHG soap, and Arm 4) all receive nasal alcohol gel the day of surgery plus two pre op showers with CHG soap.

The primary efficacy outcome will be eradication of SA colonization at all 5 body sites. Secondary outcomes will be SA surgical site infections (SSIs), all SSIs, and SA healthcare associated infections (HAIs). The study will also compare eradication of SA from each of the 5 body sites as a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participanst are outpatients in orthopedic, urology, neuro, otolaryngology, plastic and general surgery and OB/GYN clinics who are scheduled to undergo surgery at participating trial sites.
* Anticipated surgery ≥ 10 days after the date of enrollment, to allow time for completion of baseline cultures and the decolonization protocol.
* Age ≥ 18 years
* Ability to complete the decolonization protocol pre-operatively as an outpatient.
* No antibiotic therapy at the time of, or seven days prior to, baseline cultures, and no subsequent antibiotic therapy prior to the surgical procedure. Standard pre-op antibiotic prophylaxis given.
* Patients are having skin incisions as part of their scheduled surgical procedure.

Exclusion Criteria:

* Inability to give informed consent
* Surgery anticipated <10 days after the baseline cultures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will recruit patients from outpatient surgical clinics at the time their surgical procedures are planned. The study team will work with collaborating surgeons at UMMC to identify these patients. The study will recruit the following NIH priority populations: low income groups, minority groups, women, the elderly and individuals with special health care needs, including individuals with disabilities and individuals who need chronic care. These patients will be part of the surgical clinics' patient population and will be approached to participate in the study at the time their surgery is planned with their surgeon.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy in eradicating Staphylococcus aureus (SA) | baseline
  The study will compare the efficacy of four different decolonizing approaches and products in eradicating Staphylococcus aureus (SA) before surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Kline, MD, MPH, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center and Clinics, Minneapolis, Minnesota, United States